CLINICAL TRIAL: NCT05611827
Title: Comparing the Pharmacological Profile of Different Quercetin Formulations in Healthy Volunteers
Brief Title: Pharmacological Profile of Different Quercetin Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03-002
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quercetin LipoMicel (250 mg) (Experimental): Each participant receives their treatment of Quercetin LipoMicel at a total dose of 250 mg quercetin. Treatments are consumed with a glass of water (approx. 200 mL), but with no food (4hr fasting condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24hrs following a single-dose administration of quercetin and at 25, 47, 48, 71 and 72hrs after a repeated oral total dose of 250 mg LipoMicel (once daily for 72hrs). A washout period of at least 7 days between each treatment will be used.
  Interventions: Dietary Supplement: Quercetin LipoMicel (250 mg)
- Quercetin LipoMicel (500 mg) (Experimental): Each participant receives their treatment of Quercetin LipoMicel at a total dose of 500 mg quercetin. Treatments are consumed with a glass of water (approx. 200 mL), but with no food (4hr fasting condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24hrs following a single-dose administration of quercetin and at 25, 47, 48, 71 and 72hrs after a repeated oral total dose of 500 mg LipoMicel (once daily for 72hrs). A washout period of at least 7 days between each treatment will be used.
  Interventions: Dietary Supplement: Quercetin LipoMicel (500 mg)
- Quercetin LipoMicel (1000 mg) (Experimental): Each participant receives their treatment of Quercetin LipoMicel at a total dose of 1000 mg quercetin. Treatments are consumed with a glass of water (approx. 200 mL), but with no food (4hr fasting condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24hrs following a single-dose administration of quercetin and at 25, 47, 48, 71 and 72hrs after a repeated oral total dose of 1000 mg LipoMicel (once daily for 72hrs). A washout period of at least 7 days between each treatment will be used.
  Interventions: Dietary Supplement: Quercetin LipoMicel (1000 mg)
- Regular/standard Quercetin (500 mg) (Experimental): Each participant receives their treatment of standard/raw Quercetin at a total dose of 500 mg quercetin. Treatments are consumed with a glass of water (approx. 200 mL), but with no food (4hr fasting condition). A standardized lunch and dinner are served after 4h and 8h of product administration. Capillary whole blood samples are collected (after a 10hr overnight fast) at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 24hrs following a single-dose administration of quercetin. A washout period of at least 7 days between each treatment will be used.
  Interventions: Dietary Supplement: Regular/standard Quercetin (500 mg)

INTERVENTIONS:
Dietary Supplement: Quercetin LipoMicel (250 mg) — Quercetin LipoMicel® soft-gels. Total dose of 250 mg of quercetin
  Arms: Quercetin LipoMicel (250 mg)
Dietary Supplement: Quercetin LipoMicel (500 mg) — Quercetin LipoMicel® soft-gels. Total dose of 500 mg of quercetin
  Arms: Quercetin LipoMicel (500 mg)
Dietary Supplement: Quercetin LipoMicel (1000 mg) — Quercetin LipoMicel® soft-gels. Total dose of 1000 mg of quercetin
  Arms: Quercetin LipoMicel (1000 mg)
Dietary Supplement: Regular/standard Quercetin (500 mg) — Total dose of 500 mg of quercetin
  Arms: Regular/standard Quercetin (500 mg)

SUMMARY:
This study aims to evaluate the pharmacokinetics of quercetin in healthy participants after the administration of different formulations in a single- and multiple-dose phase. In the single-dose study, plasma uptake (AUC0-24 and Cmax) of standard quercetin is compared with that of LipoMicel®-a novel food-grade delivery form of quercetin. In the multiple dose study, accumulating plasma concentrations of formulated quercetin are observed over 72hrs, after repeated doses of LipoMicel treatments (AUC0-72).

At least ten healthy adults participate in an open-label, diet-controlled, crossover, plasma uptake study. Participants receive three different doses (250 mg, 500 mg or 1000 mg) of quercetin aglycone orally.

DETAILED DESCRIPTION:
Objective of this study is to investigate the pharmacokinetic profile of formulated quercetin (LipoMicel®), administered at three different doses, in healthy participants and compare it with that of a standard formulation. The pharmacokinetics of the different quercetin treatments are observed over 24hrs after a single orally administered dose of quercetin (e.g., using AUC0-24 and Cmax). Furthermore, the accumulating plasma concentrations of formulated quercetin are monitored over a 72hr period (e.g., using AUC0-72), following multiple orally administered doses of LipoMicel treatments (250 mg-1000 mg) plus the circulating metabolites of quercetin are determined in the human plasma.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* healthy, good physical condition

Exclusion Criteria:

* pregnancy or breast-feeding
* gastrointestinal conditions (acute or chronic)
* liver disease (acute or chronic)
* kidney disease (acute or chronic)
* cardiovascular disease (acute or chronic)
* hematological disease
* diabetes
* allergy or intolerance to gluten
* allergy or intolerance to quercetin
* use of any form of nicotine or tobacco, CBD/THC
* alcohol and substance abuse history
* use of medications (e.g., anti-inflammatory)
* use of quercetin supplements
* participation in another investigational study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To evaluate the plasma uptake of orally ingested quercetin (aglycone) in a novel formulation ("LipoMicel") in healthy adults by comparing the Area under the concentration-time curve (AUC) with that of standard/regular quercetin (aglycone).
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To evaluate the plasma uptake of orally ingested quercetin (aglycone) in a novel formulation ("LipoMicel") in healthy adults by comparing the Peak Plasma Concentration (Cmax) with that of standard/regular quercetin (aglycone).
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To evaluate the plasma uptake of orally ingested quercetin (aglycone) in a novel formulation ("LipoMicel") in healthy adults by comparing the time point of maximum plasma concentration (Tmax) with that of standard/regular quercetin (aglycone).

SECONDARY OUTCOMES:
AUC: the area under the concentration-time curve (quercetin metabolites) | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To determine the plasma concentrations of quercetin metabolites following the oral consumption of LipoMicel® 250 mg, over a period of 72hrs, by calculating AUC.
Cmax: maximum plasma concentration (quercetin metabolites) | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To determine the peak plasma concentrations of quercetin metabolites following the oral consumption of LipoMicel® 250 mg, over a period of 72hrs, by calculating Cmax.
Tmax: the time point of maximum plasma concentration (quercetin metabolites) | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours
  To determine the time point of maximum plasma concentration of quercetin metabolites following the oral consumption of LipoMicel® 250 mg, over a period of 72hrs, by calculating Tmax.

CONTACTS AND LOCATIONS:
Locations (1):
- ISURA, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solnier J, Zhang Y, Roh K, Kuo YC, Du M, Wood S, Hardy M, Gahler RJ, Chang C. A Pharmacokinetic Study of Different Quercetin Formulations in Healthy Participants: A Diet-Controlled, Crossover, Single- and Multiple-Dose Pilot Study. Evid Based Complement Alternat Med. 2023 Aug 10;2023:9727539. doi: 10.1155/2023/9727539. eCollection 2023. PMID 37600550